CLINICAL TRIAL: NCT05178264
Title: Transverse Myelitis Related to SARS-CoV-2 Vaccines in Patients: an Observational and Retrospective Study Using the WHO's Pharmacovigilance Database
Brief Title: Transverse Myelitis Related to SARS-CoV-2 Vaccines
Status: Completed | Type: Observational
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Other Study IDs: Pharmaco 20211210
Record Dates: First submitted 2022-01-03; First posted 2022-01-05 (Actual); Last update posted 2022-01-05 (Actual); Status verified 2021-12

CONDITIONS: Vaccine Adverse Reaction
MeSH Terms: interventions — COVID-19 Vaccines; BNT162 Vaccine; 2019-nCoV Vaccine mRNA-1273; Ad26COVS1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

INTERVENTIONS:
Drug: SARS-CoV-2 vaccines — All patients treated at least with 1 SARS-CoV-2 vaccine
  Other Names: (ChAdOx1nCov-19 (Oxford-AstraZeneca), BNT162b2 (Pfizer/BioNTech), mRNA-1273 (Moderna) and Ad26.COV2.S (Janssen/Johnson & Johnson))

SUMMARY:
Few patients receiving SARS-CoV-2 vaccines may experience rare but serious adverse events such as transverse myelitis (TM). Today, data about TM are scarce.

The objective was to investigate reports of TM adverse events related to SARS-CoV-2 vaccines labelled by FDA and EMA, including ChAdOx1nCov-19 (Oxford-AstraZeneca), BNT162b2 (Pfizer/BioNTech), mRNA-1273 (Moderna) and Ad26.COV2.S (Janssen/Johnson & Johnson) and using the World Health Organization's (WHO) pharmacovigilance database: VigiBase.

DETAILED DESCRIPTION:
Here, investigators use the World Health Organization's (WHO) database of individual safety case reports, to identify cases of TM related to SARS-CoV-2 vaccines.

ELIGIBILITY:
Inclusion Criteria:

- case reported in the World Health Organization (WHO) database (VigiBase) of individual safety case reports at the time of the extraction,

Exclusion Criteria:

* chronology not compatible between the SARS-CoV-2 vaccine adminisration and onset of TM.
* vaccines non-labelled by FDA/EMA (data cutoff december 10, 2021)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All patients
Sampling Method: Non-Probability Sample
Enrollment: 580 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2021-12-10 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
TM reportes related to SARS-CoV-2 vaccine | date of the first AE related to a SARS-CoV-2 vaccine to December 10, 2021

SECONDARY OUTCOMES:
Description of the latency period since SARS-CoV-2 vaccine exposure. | date of the first AE related to a SARS-CoV-2 vaccine to December 10, 2021
Description of the outcomes following TM | date of the first AE related to a SARS-CoV-2 vaccine to December 10, 2021
Description of patients who experienced co-reported adverse events | date of the first AE related to a SARS-CoV-2 vaccine to December 10, 2021

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandre Joachim, Caen, Basse Normandie, France

IPD SHARING:
Plan to Share IPD: No